CLINICAL TRIAL: NCT03348306
Title: Assessement of a Multi-organ Screening Procedure for the Detection of Pre-clinical Ischaemia in Antiphospholipid Syndrome The COBRA Study (CardiO-Brain Renal Involvement in Antiphospholipid Syndrome)
Brief Title: Multi-organ Screening for Asymptomatic Ischaemia in Antiphospholipid Syndrome
Acronym: COBRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Virginie Dufrost, Doctor, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-A02345-48
Record Dates: First submitted 2017-08-28; First posted 2017-11-20 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Antiphospholipid Syndrome
MeSH Terms: conditions — Antiphospholipid Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental)
  Interventions: Device: MRI; Biological: Blood sample collection

INTERVENTIONS:
Device: MRI — Brain and cardiac MRI in one time with gadolinium injection.
Biological: Blood sample collection — A blood sampling is also collected for hematocrit measure.

SUMMARY:
Introduction

AntiPhospholipid antibody Syndrome (APS) is an acquired autoimmune disorder defined by the presence of persistent thrombosis or obstetric manifestations together with the presence of persistent antiphospholipid antibodies (aPL). Patients are young and at high risk of recurrence. The current challenge is the identification of patients at high risk of organ damage that directly impact morbidity and mortality.

Small vessels thrombosis can be asymptomatic but detectable by MRI. Apart from APS, it was shown that the detection of asymptomatic ischemic events identify patients at risk for symptomatic ischemic events. Demonstrating this in patients with APS would prevent thrombotic complications.

The investigators' hypothesis is that a significant proportion of patients with APS would have asymptomatic organ involvement.

Objectives

The primary objective is to determine the frequency of asymptomatic target organ (s) (heart, brain, kidney) in APS patients.

Secondary objectives are (i) to determine the frequency of each type of MRI abnormality, (ii) to identify the factors associated with asymptomatic target organ lesion, (iii) to describe the parameters of echocardiography associated with cerebral and cardiac MRI, and (iv) to assess the feasibility of a one-time cardiovascular and brain MRI.

Methods and analysis

This is a prospective interventional, cross-sectional, non-randomized, monocentric clinical study. The investigators expect to include 50 consecutive patients with APS followed in the department of Vascular Medicine at Nancy University Hospital.

Within 15 days post-inclusion, a one-time cardiac and cerebral MRI will be performed. For each patient, the number of target organs involvements will be calculated and the frequencies will be compared by Fisher or chi-2 tests.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* Patients with documented primary thrombotic and / or obstetrical APS that respond to the revised Sapporo-Sydney classification criteria
* Person affiliated to a social security insurance,
* Person who have received complete information about the organization of the research and have signed informed consent,
* Person who has carried out a suitable clinical examination prior to the research.

Exclusion Criteria:

* Personal history of myocardial infarction, ischemic stroke or severe renal insufficiency,
* Patients with a contraindication to MRI: in particular implantable cardiac pacemakers or defibrillators, implanted pumps, cochlear implants, neurosurgical clips, intraorbital or brain metallic foreign material,
* Impossibility to perform the MRI examination, especially claustrophobic patients, or with a morphotype that does not allow access to MRI (abdominal diameter too large),
* Patient with a contraindication to Gadolinium injection: severe renal insufficiency, allergy to Gadolinium salts (precautions for use in patients at high risk of convulsions),
* APS associated with autoimmune disease (systemic lupus erythematosus according to American College of Rheumatology criteria),
* Patient with known microalbuminuria > 30mg/L,
* Women of childbearing age who do not have effective contraception,
* Persons referred to in Articles L. 1121-5 to L. 1121-8, L1122-2 and L. 1122-1-2 of the French Public Health Code :

  * Pregnant, parturient or nursing mother
  * Person deprived of liberty by judicial or administrative decision
  * Person undergoing psychiatric care
  * Person admitted to a health or social institution for other purposes than research
  * Minor person (not emancipated)
  * A major person under a measure of legal protection (guardianship, curator, safeguard of justice)
  * Person in an emergency situation
  * A major person who is unable to express his / her consent and is not under a juridical protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
A brain or cardiac involvement will be defined by the identification of specific criteria visible by MRI. | Through study completion, in average of 24 months
Renal damage will be defined by the identification of a microalbuminuria> 30mg / L. | Through study completion, in average of 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Virginie DUFROST, Principal Investigator — Nancy Academic Hospital
Locations (1):
- CHRU Nancy Brabois, Nancy, France